CLINICAL TRIAL: NCT07106424
Title: Liquid Biopsy for Early Screening Cohort Study of Multiple Gastrointestinal Tumors
Brief Title: Early Screening Cohort Study of Multiple Gastrointestinal Tumors
Status: Recruiting | Type: Observational
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, Academician of the Chinese Academy of Engineering, President of Shandong Cancer Hospital, Shandong Cancer Hospital and Institute
Other Study IDs: DECIPHER-GASTRO
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Early Detection of Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- gastrointestinal tumor screening: They will undergo cancer screening based on liquid biopsy as well as routine gastrointestinal endoscopy screening simultaneously.

SUMMARY:
Gastrointestinal tumors, including esophageal cancer, gastric cancer, and colorectal cancer, are among the most common and highly prevalent malignant tumors in Shandong Province. Currently, most patients seek medical attention only after clinical symptoms appear, by which time the disease has already reached an intermediate or advanced stage. This leads to increased treatment costs and poorer therapeutic outcomes. Early detection and intervention through screening are effective measures to improve the cure rate of gastrointestinal tumors and reduce their incidence and mortality rates.

This project leverages the Shandong Province Tumor Screening and Early Diagnosis & Treatment Platform and is based on the ongoing Shandong Gastrointestinal Cancer Screening Cohort. It aims to collect 4,000 plasma samples from individuals undergoing simultaneous screening for esophageal, gastric, and colorectal cancers. Using Nanjing Shihe Medical Laboratory's independently developed multi-cancer early detection liquid biopsy product for gastrointestinal cancers, the study will further validate the performance of liquid biopsy in multi-cancer screening by correlating results with endoscopic findings (gastroscopy and colonoscopy).

DETAILED DESCRIPTION:
Esophageal cancer, gastric cancer, and colorectal cancer are common gastrointestinal malignancies in China, accounting for 25.54% of all cancer cases and 33.93% of cancer-related deaths nationwide. Early detection, diagnosis, and treatment of these cancers have proven to be effective strategies for cancer prevention and control, serving as key measures to reduce mortality rates and improve survival outcomes.

Gastrointestinal tumors are also highly prevalent in our province. According to the 2022 Shandong Provincial Tumor Registry Annual Report, approximately 27,000 new cases of upper gastrointestinal cancers (including esophageal and gastric cancers) and colorectal cancer were recorded in registered areas, representing 24.71% of all malignant tumor cases. Deaths from these cancers reached about 16,300, accounting for 24.11% of all cancer-related deaths.

In recent years, with support from national public health funding, the Shandong Cancer Center has organized screening programs across the province, completing over 600,000 screenings for upper gastrointestinal and colorectal cancers. These efforts have detected more than 13,000 cases of precancerous or early-stage lesions, with a positive detection rate of 2.23%. Among these, 10,500 cases were diagnosed at an early stage, achieving an early diagnosis rate exceeding 80%, demonstrating significant societal benefits. Regions such as Feicheng, Linqu, and Dongping have established early diagnosis and treatment centers for upper gastrointestinal cancers, enabling comprehensive full-cycle management from screening to treatment and follow-up. This progress lays a crucial foundation for large-scale, long-term cohort studies.

This research is based on the ongoing Shandong Gastrointestinal Cancer Screening Cohort and will collect plasma samples from 4,000 individuals undergoing simultaneous screening for esophageal, gastric, and colorectal cancers. The study will utilize an independently developed multi-cancer early detection (MCED) liquid biopsy technology for performance validation.

ELIGIBILITY:
Inclusion Criteria:

* gastrointestinal cancer screening population
* age 40-75
* no prior history of tumors

Exclusion Criteria:

* Severe heart disease, heart failure;
* Severe respiratory disease, dyspnea, continuous asthma, or those with serious brain diseases;
* Severe spinal deformity, or patients with aneurysms;
* Physically weak and unable to tolerate endoscopy, or those who have difficulty remaining calm and self-controlled;
* Acute corrosive inflammation of the gastrointestinal tract, or those suspected of having a gastrointestinal perforation;
* Large amounts of ascites, severe abdominal distension, or severe esophageal varices;
* Those with a tendency to bleed (abnormal coagulation function), or those taking anticoagulant medications. The latter must discontinue the medication for one week and have normal coagulation function before undergoing endoscopy;
* Pregnant women;
* Those with a history of iodine allergy, etc.
* Patients who have been diagnosed with tumors or have a history of prior tumors.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals undergoing screening for esophageal cancer, gastric cancer, and colorectal cancer within the Shandong Province gastrointestinal screening cohort aged 40-74 years.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2028-09-10 (Estimated); Study Completion 2030-09-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity for detection of high-grade (or above) gastric/esophageal/colorectal cancer | 2024.7-2027.7
  Primary Objective:
  Sensitivity for detecting high-grade or above gastric/esophageal/colorectal lesions.
  Secondary Objectives:
  Positive predictive value (PPV), specificity, and negative predictive value (NPV) for detecting high-grade or above gastric/esophageal/colorectal lesions.
  PPV and sensitivity for detecting other cancer types.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided
The data sharing plan is pending final approval by the institutional review board (IRB) and sponsor. A decision will be made prior to manuscript submission to journals

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/40571756/